CLINICAL TRIAL: NCT05015868
Title: Contribution of Genetics, Non-invasive Neurophysiological Methods, Neuroimaging and Neuropsychology in Identifying the Cause and the Epileptogenic Zone in Focal Cryptogenic Epilepsies
Brief Title: Contribution of Genetics, Non-invasive Methods and Neuropsychology in Focal Cryptogenic Epilepsies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 879
Record Dates: First submitted 2021-08-11; First posted 2021-08-20 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Epilepsies, Partial; Epilepsy Intractable
MeSH Terms: conditions — Epilepsies, Partial; Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IDENTIFICATION OF THE CAUSE OF THE EPILEPSY AND OF THE EPILEPTOGENIC ZONE (sequential approach) (Experimental): Step1: standard of care.
  * acquisition and updating of Electroencephalogram polygraphic data of wakefulness and sleep and neuroradiological data
  * complete neuropsychological assessment
  * genetic tests through Next generation sequencing epilepsies panel, or exome
  Step 2: experimental
  - combined Electroencephalogram-Functional brain magnetic resonance imaging registration.
  Step 3: experimental
  In the event that neither the cause nor the epileptogenic area has been identified, we will evaluate the execution of further tests, such as:
  * execution of High Density-Electroencephalogram recording at "IRCCS Medea di Conegliano" (TV, Italy) (approximately 3 patients / year) for a further electrophysiological definition;
  * 7 Tesla brain magnetic resonance imaging performed at "IRCCS Stella Maris in Calambrone"(PI, Italy) (approximately 3 patients / year expected), to obtain greater spatial resolution and better neuroradiological definition.
  Interventions: Diagnostic Test: Standard of care; Diagnostic Test: Functional magnetic resonance imaging-Electroencephalogram combined analysis; Diagnostic Test: High density- electroencephalogram or 7 Tesla magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Standard of care — Enrollment of patients afferent to our Center with cryptogenic drug-resistant epilepsy with onset in pediatric age, subject to informed consent;
  * acquisition and updating of Electroencephalogram polygraphic data of wakefulness and sleep and neuroradiological data (previous negative brain magnetic resonance imaging);
  * execution of a complete neuropsychological assessment for the classification of cognitive aspects and evaluation of executive functions;
  * execution of genetic tests through Next generation sequencing epilepsies panel or exome sequencing
Diagnostic Test: Functional magnetic resonance imaging-Electroencephalogram combined analysis — A functional brain magnetic resonance imaging is executed analysing blood oxygenation level dependent signal.
  During the functional recording, a contemporary electroencephalogram is registered in order to analyse the space-time relationship between the epileptic discharges and the bold abnormalities.
Diagnostic Test: High density- electroencephalogram or 7 Tesla magnetic resonance imaging — In the event that neither the cause nor the epileptogenic area has been identified, we will evaluate the execution of further tests, such as:
  * execution of High Density-electroencephalogram recording at "IRCCS Medea di Conegliano" (TV, Italy) (approximately 3 patients / year) for a further electrophysiological definition;
  * 7 Tesla brain magnetic resonance imaging performed at "IRCCS Stella Maris in Calambrone" (PI, italy) (approximately 3 patients / year expected), to obtain greater spatial resolution and better neuroradiological definition.

SUMMARY:
Patients with cryptogenic focal epilepsy (unknown cause) represent about the 30% of the entire population of epilepsy patients. Among them, about 30% are drug-resistant. The implementation of of high-field magnetic resonance imaging resolution, the new Next Generation Sequencing techniques,and innovative non-invasive neurophysiological methods (Electroencephalogram-Functional magnetic resonance imaging and High Density-Electroencephalogram) could provide a superior identification of the epileptogenic zone and therefore an increased access to epilepsy surgery.

Despite this, patients with cryptogenic epilepsy require more frequently invasive methods of presurgical study and they have more unfavorable results than patients with lesions detectable on magnetic resonance imaging. Within this context, the study is aimed at integrating the neurophysiological, radiological, neuropsychological and genetic aspects of patients with focal cryptogenic epilepsy in order to evaluate their surgical eligibility,sparing invasive methods.

DETAILED DESCRIPTION:
The investigators foresee study duration of 36 months and the enrollment of about 20-25 patients, affected by cryptogenic epilepsy with onset during pediatric age (0-18 years), not only to identify the cause of epilepsy and the epileptogenic zone, but also to define in a non-invasive manner, the patient's possible eligibility for surgical therapy.

Innovative neurophysiological methods, such as combined Electroencephalogram-Functional magnetic resonance imaging recording and high resolution electroencephalogram, in addition to 7 Tesla brain magnetic resonance imaging (available through the Imago7 non-profit foundation), neuropsychological studies and genetic tests through Next generation sequencing allow an advanced pre-surgical study free from the risks and discomforts caused by invasive methods. The systematic use of these diagnostic approaches will implement the knowledge and skills of the teams and it will stimulate their use in the clinical daily practise, especially for pediatric patients.

In addition to that, the investigators would like to analyse descriptive indications relating to the diagnostic sensitivity of the combined Electroencephalogram-Functional magnetic resonance imaging recording, High Density-electroencephalogram and 7 Tesla magnetic resonance imaging in the identification of the epileptogenic zone, in patients with cryptogenic focal epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* focal epilepsy, onset during pediatric age (<18 y)
* drug resistance
* unknown cause
* Brain magnetic resonance imaging negative

Exclusion Criteria:

* epilepsy with good therapeutic control
* focal symptomatic epilepsy
* age limits onset (> 18 y)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of the epileptogenic zone. | through study completion, an average of 1 year
  Identification of the epileptogenic zone. Identification of non-invasive methods (Electroencephalogram-Functional magnetic resonance imaging, High Density-Electroencephalogram and 7 Tesla brain magnetic resonance imaging) in order to provide the necessary and crucial data, allowing the patient access to the epilepsy surgery without recurring to invasive methods. The calculation of the sample size was carried out on the basis of the primary objective of non-invasive identification of the epileptogenic zone. 60 patients will be sufficient to estimate the proportion of subjects treated with an effect size of 0.5, a power of 90% and a first type error of 5%. (60 patients are obtained by including patients from Conegliano).

SECONDARY OUTCOMES:
Diagnostic sensitivity comparison | through study completion, an average of 1 year
  Diagnostic sensitivity comparison between combined Electroencephalogram-Functional magnetic resonance imaging and High Density-Electroencephalogram or 7Tesla brain magnetic resonance imaging recording for a patients subgroup.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Zambrano, MD, Principal Investigator — Scientific Institute IRCCS Eugenio Medea
Locations (1):
- Scientific Institute IRCCS Eugenio Medea, Bosisio Parini, lecco, Italy